CLINICAL TRIAL: NCT03068585
Title: Phase 3 Study of Efficiency, Safety and Portability of Gene Therapy Drug Neovasculgen (DNA Encoding the 165-amino-acid Isoform of Human Vascular Endothelial Growth Factor (pCMV - VEGF165) for Peripheral Arterial Disease Complex Treatment
Brief Title: Efficiency, Safety and Portability of Neovasculgen
Acronym: Neovasculgen
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Artgen Biotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVG-IC
Record Dates: First submitted 2011-06-14; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2011-06

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; CLI; stage 2a-3 of Pokrovsky-Fonteine
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neovasculgen (Experimental): DNA encoding the 165-amino-acid isoform of human vascular endothelial growth factor (pCMV - VEGF165)
  Interventions: Drug: Neovasculgen (Cambiogeneplasmid)
- Control (No Intervention): Control therapy

INTERVENTIONS:
Drug: Neovasculgen (Cambiogeneplasmid) — treatment
  Other Names: Neovasculgen
  Arms: Neovasculgen

SUMMARY:
In 2010, we completed a phase 1 to 2a clinical trial of pCMV-vegf165 in patients with chronic lower limb ischemia (stage 2a to 3 according to Fontaine classification modified by A. V. Pokrovsky) who were not suitable for reconstructive surgery or endovascular treatment. This study demonstrated the safety, feasibility, and short-term(3 months) efficacy of pCMV-vegf165 gene transfer,12,13which lead to conducting a phase 2b to 3 multicenter clinical trial. The study was conducted under the control of the Russian Ministry of Health and was completed in 2011. Patients enrolled in the study were subjected to a 6-month

DETAILED DESCRIPTION:
We conducted a phase 2b/3 multicenter randomized controlled clinical trial of the intramuscular transfer of a plasmid DNA encoding vascular endothelial growth factor (VEGF) 165 with cytomegalovirus promotor (CMV) in patients with atherosclerotic lower limb ischemia. A total of 100 patients were enrolled in the study, that is, 75 patients were randomized into the test group and received 2 intramuscular injections of 1.2 mg of pCMV- vegf165, 14 days apart together with standard pharmacological treatment. In all, 25 patients were randomized into the control group and received standard treatment only. The following end points were evaluated within the first 6 months of the study and during a 1.5-year additional follow-up period: pain-free walking distance (PWD), ankle-brachial index (ABI), and blood flow velocity (BFV).

ELIGIBILITY:
Inclusion Criteria:

* age more than 40 years;
* a history of stable claudication for at least 3 months;
* stage 2 to 3 chronic ischemia according to Fontaine classification (modified by A. V. Pokrovsky);
* presence of hemodynamically significant (stenosis >70% and/or occlusion) diffuse lesions of the interior and (or) posterior tibial arteries (distal lesion);
* voluntary informed consent signed and dated by the patient.

Exclusion Criteria:

* chronic lower limb ischemia of nonatherosclerotic genesis; stage 4 chronic ischemia according to Fontaine classification modified by A. V. Pokrovsky (ischemic ulcers and necrotic lesions);
* severe concomitant pathology with life expectancy <1 year;
* infectious diseases, history of cancer, or suspected malignancy;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Pain-free walking distance. | 6 months
  The PWD was determined using a treadmill test with reduced initial speed (1 km/h), as the majority of elderly patients were unable to perform Gardner test or its equivalents.

SECONDARY OUTCOMES:
Ankle-brachial index | 6 months
  The ankle-brachial pressure index (ABPI) or ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium). Compared to the arm, lower blood pressure in the leg is an indication of blocked arteries due to peripheral artery disease (PAD).
Transcutaneous oximetry | 6 months
  Transcutaneous oximetry, tcpO2 or TCOM, is a local, non-invasive measurement reflecting the amount of O2 that has diffused from the capillaries, through the epidermis.
quality of life | 6 months
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized by managed care organizations and by Medicare for routine monitoring and assessment of care outcomes in adult patients.

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Russian National Surgery Center by Petrovsky, Moscow, Central Russia
  - Ryazansky State Medical University, Ryazan, Central Russia
  - Yaroslavl State Medical Academy, Yaroslavl, Central Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deev RV, Bozo IY, Mzhavanadze ND, Voronov DA, Gavrilenko AV, Chervyakov YV, Staroverov IN, Kalinin RE, Shvalb PG, Isaev AA. pCMV-vegf165 Intramuscular Gene Transfer is an Effective Method of Treatment for Patients With Chronic Lower Limb Ischemia. J Cardiovasc Pharmacol Ther. 2015 Sep;20(5):473-82. doi: 10.1177/1074248415574336. Epub 2015 Mar 13. PMID 25770117
- [Derived] Deev R, Plaksa I, Bozo I, Mzhavanadze N, Suchkov I, Chervyakov Y, Staroverov I, Kalinin R, Isaev A. Results of 5-year follow-up study in patients with peripheral artery disease treated with PL-VEGF165 for intermittent claudication. Ther Adv Cardiovasc Dis. 2018 Sep;12(9):237-246. doi: 10.1177/1753944718786926. Epub 2018 Jul 11. PMID 29996720